CLINICAL TRIAL: NCT06688669
Title: Examining the Effects of Removable Denture on Behavior and Cognitive Skills in Geriatric Patients
Brief Title: Examining the Effects of Removable Denture Use in Patients Over 60 Years of Age
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Berk Bilgen, PhD DDS, Principal Investigator, Istanbul University
Other Study IDs: 2024/47/Rev-1
Record Dates: First submitted 2024-11-10; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Edentulism; Denture, Complete; Denture, Partial, Removable
Keywords: complete denture; removable partial denture; OHIP-14; mini mental state examination
MeSH Terms: interventions — Denture, Partial, Removable

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with complete denture: Patients with total edentulism who require complete dentures.
  Interventions: Other: Fabrication of suitable complete or removable partial dentures for the patient
- Patients with removable partial dentures: Patients with partial edentulism who require removable-partial dentures.
  Interventions: Other: Fabrication of suitable complete or removable partial dentures for the patient

INTERVENTIONS:
Other: Fabrication of suitable complete or removable partial dentures for the patient — Fabrication of suitable complete and partial dentures for the patient. The study will not interfere with this treatment process; only follow-up assessments will be conducted at specific intervals after the dentures are fabricated, and surveys will be administered to the patient.

SUMMARY:
Patients over the age of 60 who do not currently have any removable dentures but require them will be included in the study. Patients who will receive complete dentures and those who will receive partial dentures will be assessed in separate groups. Before the fabrication of the dentures, the Mini-Mental State Examination Test (MMSE), the physical normative value test (TUG), and the Oral Functional Capacity (OFC) scoring will be conducted. No intervention will be made to the treatment during the prosthetic treatment process.

The same questionnaires will be administered again three weeks after the completion of the prosthetic treatments. The impact of the use of removable dentures on test results will be evaluated. Additionally, during this session, patients will complete a patient satisfaction test regarding their dentures (OHIP-14 for patients with a removable partial denture indication, and OHIP-edent for patients with a complete denture indication). Patients will be called back after three months, and all tests will be repeated. The relationship between the Mini-Mental State Examination, the TUG test, and the OFC test with patient satisfaction will be assessed and any changes in test scores related to denture use will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 60
* No systemic condition that would prevent the fabrication of removable dentures
* Need for new removable dentures for both jaws
* Ability to read and understand the questions in the tests and surveys
* No barriers to communication or self-expression
* No significant physical disability affecting functionality
* No history of cancer or surgical operation in the head and neck region
* No conditions or medications that could limit test performance (e.g., Parkinson's disease)

Exclusion Criteria:

* Patients under the age of 60
* Patients who do not require new removable dentures
* Patients whose missing teeth can be restored with fixed prosthetic restorations and who do not need removable dentures
* Patients who are illiterate
* Patients with systemic conditions that prevent the fabrication of removable dentures
* Patients with conditions like Parkinson's disease that could restrict test performance or who use medications with side effects causing unwanted convulsions
* Patients with significant balance issues, who frequently lose balance while walking
* Geriatric patients with temporary or permanent memory loss
* Patients with any history of cancer in the head and neck region
* Patients with severe difficulty in communication and self-expression
* Patients who are not willing to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 60 who apply to Istanbul University Faculty of Dentistry to receive removable dentures.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of mini mental state examination (MMSE) test, in individuals after the use of dentures | From enrollment to three months after
  Evaluation of the effects of complete dentures and removable partial dentures on patients' cognitive status using the Mini-Mental State Examination (MMSE) test. Patients will first undergo the 10-question Mini Mental State Examination (MMSE) test. The Mini Mental State Examination assesses cognitive status by measuring verbal fluency, executive functions, and visuospatial skills. This test will evaluate the cognitive condition of the patient. The MMSE is a brief, 10-question test that takes approximately 5 minutes to complete. It will be administered through a question-and-answer format. A total score will be calculated, and statistical analysis will be conducted based on this total score. An increase in the score will indicate an improvement in cognitive status.
Evaluation of Timed up and go (TUG) test in individuals after the use of dentures | From enrollment to three months after
  Evaluation of the effects of complete dentures and removable partial dentures on patients' dynamic functions using the Timed Up and Go (TUG) test.

SECONDARY OUTCOMES:
Adaptation of dentures in geriatric patients | From enrollment to three months after
  Examining the changes in geriatric patients' adaptation to their new dentures over time and correlating their adaptation (OHIP-14 results) with their cognitive or functional status before treatment.The OHIP-14 test is frequently used to assess satisfaction with removable dentures. Based on the answers to the questions in this test, patient satisfaction is scored, with higher scores indicating greater satisfaction.
Evaluation of Oral Functional Capacity (OFC) in individuals after the use of dentures | From enrollment to three months after
  Evaluation of the effects of dentures on on patients' oral functional capacities (OFC).The OFC assessment is conducted as follows: Parameters under the titles of therapeutic capacity, oral hygiene ability, and self-responsibility are evaluated by the clinician and rated as 'reduced,' 'significantly reduced,' 'normal,' or 'absent,' with a score out of 4. Since the evaluation is conducted by the clinician, it does not present any additional challenge to the patients and takes approximately 5 minutes. Two researchers will independently assign an OFC score based on the patient's responses, aiming for consistency between the two scores. This scoring method has been used in all studies conducted with OFC (each category will be scored separately out of 4, and the average of the three scores will be taken). The results of the three tests will be evaluated through separate statistical analyses."

CONTACTS AND LOCATIONS:
Overall Officials: Olcay Şakar, Prof. Dr. Clinical Professor, Study Chair — Istanbul University
Locations (1):
- Istanbul University Faculty of Dentistry, Istanbul, Vezneciler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmed SE, Raju R, Kurien A, M K, Bano S, Shalma H. Impact of Denture Prostheses on Cognitive Functioning in Completely Edentulous Patients: A Pilot Study. Cureus. 2023 Aug 16;15(8):e43570. doi: 10.7759/cureus.43570. eCollection 2023 Aug. PMID 37719519